CLINICAL TRIAL: NCT02887261
Title: Study on Indications of "Bard" PowerPort Isp Implantable Port: Image Accuracy in Resectable Esophageal Cancer Patients
Brief Title: Study on Indications of "Bard" PowerPort Isp Implantable Port
Acronym: BPIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CGMH-IRB-104-3143A3
Record Dates: First submitted 2016-06-29; First posted 2016-09-02 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2018-12

CONDITIONS: Power Port; Image Accuracy
Keywords: Power Port

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Power Port (Other): patients who received power injectable port
  Interventions: Device: "Bard"PowerPort sip Implantable Port
- Conventional Port (Active Comparator): patients who received conventional port ( not power injectable)
  Interventions: Device: Conventional Port

INTERVENTIONS:
Device: "Bard"PowerPort sip Implantable Port — capable for power injection for contrast media.
  Arms: Power Port
Device: Conventional Port — not for power injection for contrast media.
  Arms: Conventional Port

SUMMARY:
For esophageal cancer patients,chest CT could provide more accurate staging information and eliminated operation that could not achieve R0 resection such as T4 disease. However, the variation image quality was usual encountered because of contrast medium was injected via peripheral vein. Power injectable port could provide a secure vascular access as administration route for contrast medium via central vein. This could provide higher intravascular contrast medium concentration and could lead better image quality. This study divided into two arms, one group planned to receive power injectable port and another received conventional port. The aim of study was tried to identified the image differences between different contrast medium administration route and the its survival impact of esophageal cancer.

DETAILED DESCRIPTION:
It is extremely important for cancer patients to have a reliable vascular access which may be used for administering irritant infusions, such as chemotherapeutic agents and intravenous nutrition supplement, and for drawing blood for routine examinations in the long term. To address patients' needs, Aubaniac introduced the central vein puncture technique for vascular infusion in 1952AD. With this technique, patients were allowed to take intravenous infusion safely but had to experience repeated punctures every 5-7 days for preventing tunnel tract infection. Later, with the improvement of medical material, the first indwelling intravenous catheter was designed by BrovIac which could be implanted for a period of time. In 1979, based on this prototype, Hickmen added a subcutaneous cuff in order to separate the proximal part of catheter from environment and minimize the risk of tunnel tract infusion, leading to cosmetic concerns and compromising patients' daily activities . It's till 1982 that Dr. Niederhuber developed the totally implantable venous device, which made vascular access set up simpler for patients. However, low injection pressure setting constrained some applications, such as power injection of contrast media for CT scan. Therefore, peripheral venous puncture was still inevitable sometimes for the patients with intravenous access devices placed.

Patients with cancer need to regularly receive imaging surveillance to evaluate treatment efficacy. Besides, the surveillance imaging provides benchmark reference for adjustment of treatment plan. To provide the enhanced quality of image, contrast media is expected to be administered at certain injection rates. Such requested injection rates would generate high pressures due to the sticky nature of the contrast media. Most of the time, the pressures incurred are far beyond the pressure setting of the conventional ports which mostly in the range of 10 ~ 12 atmospheric pressures (approximately 145 ~ 175 psi) and may cause device rupture or burst. Venipuncture is still unavoidable for oncologic patients with intravenous port implanted for administering contrast media so that patients' vessels cannot be completely protected from repeated venipunctures. Besides, patients' native vessel has its own infusion pressure limitation. Extravasation of contrast media to peripheral soft tissues would happen to the patients with poor vessels or to those in need for power injection of contrast media. Extravasation of contrast media may lead to cutaneous necrosis at different degrees. Such a consequence not only causes pain to patients, but also postpones the subsequent treatment that cannot be continued until the wound is healed up. The delay of treatment might impact on patients' survival. To avoid such a complication, radiologists are forced to lower the infusion velocity of contrast media and compromise the quality of the image requested by the diagnosis.

Tumor would induce neovascularization process which may trigger abnormal new vessels to form and surround the lesion for providing the requested nutritional support for its growth. Given by this characteristic, the contrast-enhanced image plays an important role in evaluating the degree of tumor invasion. In addition, information regarding relative anatomic relationship between tumor and surrounding vital structure is also crucial for formulation of a treatment plan. However, as medical image is not color but black and white images, images with sharp contrast can present subtle changes of tumor more clearly as reference for evaluation of physicians. If the resectability and the metastatic lesions could be identified from medical images as early as possible, personalized treatment could be planned to achieve better survival rates. Therefore, it is extremely important to acquire a clear medical image. With respect to conventional CT, it can indicate the relative anatomical relationship between tumor and surrounding vital structures, which is a key basis for formulation of treatment plan. Current initial imaging data shows CT images taken after infusion with an implanted port that can endure a high infusion pressure are actually different from those taken after infusion through peripheral vein Theoretically, contrast media administrated via central vein could increase concentration of contrast media within a short time, improving the imaging quality of tissues close to the tumor greatly and reducing the necessity of peripheral venipuncture and the risk of contrast extravasation. Therefore, an implantable port that can endure a high infusion pressure is the only solution to meet the demand both from treatment and from surveillance. Furthermore, venous thrombus is more likely to occur in patients with malignant tumor, which must be prevented as it may cause a higher in-hospital mortality rate. If loosen thrombus delivered by venous return may lead most serious complications, such as pulmonary embolism. Pulmonary artery angiography was used to be the only way for diagnosis. However, with the improvement of imaging technology, computed tomography now could be utilized in diagnosis too. High quality of image may be achieved as long as contrast media is injected at a high velocity but patients might risk getting hurt by extravasation of contrast media. After intravenous port that could endure high injection pressure was available, the characteristic of high volume profile could provide secure vascular route with minimal risk of extravasation. However, there was no agreeable conclusion on how such a device may benefit the survival of the patients. Although the port that can endure a high pressure of infusion can provide a reliable intravenous route and better medical images, the benefits of prognosis which may be brought by such port are still unknown. Besides, the national insurance hasn't reimbursed such new type of infusion port due to limited insurance budget. Therefore, investigators intend to identify the patients suitable for implantation of such port in view of features of imaging and tumor so as to improve prognosis of cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with esophageal cancer that in the clinical stage of T3~4 N0~2 M0 before treatment and presents no distant metastasis

Exclusion Criteria:

* Patients with esophageal cancer that in the clinical stage of TxN3M1 before treatment and presents no distant metastasis

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-05; Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Chest tomography (Before and after neoadjuvant therapy) | 1. before neoadjuvant CCRT ( just after diagnosis) 2. after neoadjuvant CCRT prior surgery intervention(for treatment response after neoadjuvant CCRT; 3~4 months after neoadjuvant CCRT.)
  tumor invasion status ( CT result)
endoscopic ultrasound (Before and after neoadjuvant therapy) | 1. before neoadjuvant CCRT ( just after diagnosis) 2. after neoadjuvant CCRT prior surgery intervention(for treatment response after neoadjuvant CCRT; 3~4 months after neoadjuvant CCRT.)
  tumor invasion status ( EBUS image result)
pathologic report | After curative surgery ( 3-4 months after treatment completion)
  Real tumor invasion status

SECONDARY OUTCOMES:
Chest tomography (Before and after neoadjuvant therapy) | 1. before neoadjuvant CCRT ( just after diagnosis) 2. after neoadjuvant CCRT prior surgery intervention( 3-4 months after neoadjuvant CCRT)
  Tumor size shrinkage

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Yang Wu, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Charvat J, Linke Z, Horaekova M, Prausova J. Implantation of central venous ports with catheter insertion via the right internal jugular vein in oncology patients: single center experience. Support Care Cancer. 2006 Nov;14(11):1162-5. doi: 10.1007/s00520-006-0073-2. Epub 2006 Apr 5. PMID 16596418
- [Background] Copper CM, Pacanowski JP, Bell JL. The trapezius port: a novel approach for port access. Am Surg. 2005 Feb;71(2):106-9. PMID 16022007
- [Background] Broviac JW, Cole JJ, Scribner BH. A silicone rubber atrial catheter for prolonged parenteral alimentation. Surg Gynecol Obstet. 1973 Apr;136(4):602-6. No abstract available. PMID 4632149
- [Background] Hickman RO, Buckner CD, Clift RA, Sanders JE, Stewart P, Thomas ED. A modified right atrial catheter for access to the venous system in marrow transplant recipients. Surg Gynecol Obstet. 1979 Jun;148(6):871-5. No abstract available. PMID 109934
- [Background] Niederhuber JE, Ensminger W, Gyves JW, Liepman M, Doan K, Cozzi E. Totally implanted venous and arterial access system to replace external catheters in cancer treatment. Surgery. 1982 Oct;92(4):706-12. PMID 7123491
- [Background] Belzunegui T, Louis CJ, Torrededia L, Oteiza J. Extravasation of radiographic contrast material and compartment syndrome in the hand: a case report. Scand J Trauma Resusc Emerg Med. 2011 Feb 4;19:9. doi: 10.1186/1757-7241-19-9. PMID 21294896
- [Background] Azais H, Bresson L, Bassil A, Katdare N, Merlot B, Houpeau JL, El Bedoui S, Meurant JP, Tresch E, Narducci F. Chemotherapy drug extravasation in totally implantable venous access port systems: how effective is early surgical lavage? J Vasc Access. 2015 Jan-Feb;16(1):31-7. doi: 10.5301/jva.5000316. Epub 2014 Oct 16. PMID 25362986
- [Background] Petterson TM, Marks RS, Ashrani AA, Bailey KR, Heit JA. Risk of site-specific cancer in incident venous thromboembolism: a population-based study. Thromb Res. 2015 Mar;135(3):472-8. doi: 10.1016/j.thromres.2014.12.013. Epub 2014 Dec 16. PMID 25547213
- [Background] Lyman GH, Bohlke K, Khorana AA, Kuderer NM, Lee AY, Arcelus JI, Balaban EP, Clarke JM, Flowers CR, Francis CW, Gates LE, Kakkar AK, Key NS, Levine MN, Liebman HA, Tempero MA, Wong SL, Somerfield MR, Falanga A; American Society of Clinical Oncology. Venous thromboembolism prophylaxis and treatment in patients with cancer: american society of clinical oncology clinical practice guideline update 2014. J Clin Oncol. 2015 Feb 20;33(6):654-6. doi: 10.1200/JCO.2014.59.7351. Epub 2015 Jan 20. PMID 25605844
- [Background] Baptista R, Santiago I, Jorge E, Teixeira R, Mendes P, Curvo-Semedo L, Castro G, Monteiro P, Caseiro-Alves F, Providencia LA. One-shot diagnostic and prognostic assessment in intermediate- to high-risk acute pulmonary embolism: the role of multidetector computed tomography. Rev Port Cardiol. 2013 Jan;32(1):7-13. doi: 10.1016/j.repc.2012.05.020. Epub 2012 Dec 11. PMID 23245344
- [Background] Rice TW. Clinical staging of esophageal carcinoma. CT, EUS, and PET. Chest Surg Clin N Am. 2000 Aug;10(3):471-85. PMID 10967751
- [Background] Sandha GS, Severin D, Postema E, McEwan A, Stewart K. Is positron emission tomography useful in locoregional staging of esophageal cancer? Results of a multidisciplinary initiative comparing CT, positron emission tomography, and EUS. Gastrointest Endosc. 2008 Mar;67(3):402-9. doi: 10.1016/j.gie.2007.09.006. PMID 18178202
- [Background] Sloof GW. Response monitoring of neoadjuvant therapy using CT, EUS, and FDG-PET. Best Pract Res Clin Gastroenterol. 2006;20(5):941-57. doi: 10.1016/j.bpg.2006.04.004. PMID 16997171
- [Background] Yegin EG, Duman DG. Staging of esophageal and gastric cancer in 2014. Minerva Med. 2014 Oct;105(5):391-411. Epub 2014 Jul 7. PMID 25000218
- [Background] Isenberg G, Chak A, Canto MI, Levitan N, Clayman J, Pollack BJ, Sivak MV Jr. Endoscopic ultrasound in restaging of esophageal cancer after neoadjuvant chemoradiation. Gastrointest Endosc. 1998 Aug;48(2):158-63. doi: 10.1016/s0016-5107(98)70157-9. PMID 9717781
- [Background] Li SH, Rau KM, Lu HI, Wang YM, Tien WY, Liang JL, Lin WC. Pre-treatment maximal oesophageal wall thickness is independently associated with response to chemoradiotherapy in patients with T3-4 oesophageal squamous cell carcinoma. Eur J Cardiothorac Surg. 2012 Dec;42(6):958-64. doi: 10.1093/ejcts/ezs136. Epub 2012 Mar 30. PMID 22466694
- [Background] Teichgraber UK, Gebauer B, Benter T, Wagner HJ. Central venous access catheters: radiological management of complications. Cardiovasc Intervent Radiol. 2003 Jul-Aug;26(4):321-33. doi: 10.1007/s00270-003-0112-z. PMID 14667113
- [Background] Steuer CE, Behera M, Kim S, Patel N, Chen Z, Pillai R, Saba NF, Shin DM, Owonikoko TK, Khuri FR, Ramalingam SS. Predictors and outcomes of venous thromboembolism in hospitalized lung cancer patients: A Nationwide Inpatient Sample database analysis. Lung Cancer. 2015 Apr;88(1):80-4. doi: 10.1016/j.lungcan.2015.01.022. Epub 2015 Feb 2. PMID 25726042
- [Background] Wani S, Das A, Rastogi A, Drahos J, Ricker W, Parsons R, Bansal A, Yen R, Hosford L, Jankowski M, Sharma P, Cook MB. Endoscopic ultrasonography in esophageal cancer leads to improved survival rates: results from a population-based study. Cancer. 2015 Jan 15;121(2):194-201. doi: 10.1002/cncr.29043. Epub 2014 Sep 18. PMID 25236485
- [Background] Yen TJ, Chung CS, Wu YW, Yen RF, Cheng MF, Lee JM, Hsu CH, Chang YL, Wang HP. Comparative study between endoscopic ultrasonography and positron emission tomography-computed tomography in staging patients with esophageal squamous cell carcinoma. Dis Esophagus. 2012 Jan;25(1):40-7. doi: 10.1111/j.1442-2050.2011.01204.x. Epub 2011 May 19. PMID 21595776
- [Background] Cerfolio RJ, Bryant AS, Ohja B, Bartolucci AA, Eloubeidi MA. The accuracy of endoscopic ultrasonography with fine-needle aspiration, integrated positron emission tomography with computed tomography, and computed tomography in restaging patients with esophageal cancer after neoadjuvant chemoradiotherapy. J Thorac Cardiovasc Surg. 2005 Jun;129(6):1232-41. doi: 10.1016/j.jtcvs.2004.12.042. PMID 15942562
- [Background] Pfau PR, Perlman SB, Stanko P, Frick TJ, Gopal DV, Said A, Zhang Z, Weigel T. The role and clinical value of EUS in a multimodality esophageal carcinoma staging program with CT and positron emission tomography. Gastrointest Endosc. 2007 Mar;65(3):377-84. doi: 10.1016/j.gie.2006.12.015. PMID 17321235
- [Background] Kalha I, Kaw M, Fukami N, Patel M, Singh S, Gagneja H, Cohen D, Morris J. The accuracy of endoscopic ultrasound for restaging esophageal carcinoma after chemoradiation therapy. Cancer. 2004 Sep 1;101(5):940-7. doi: 10.1002/cncr.20429. PMID 15329901
- [Background] van den Hoed RD, Feldberg MA, van Leeuwen MS, van Dalen T, Obertop H, Kooyman CD, van der Schouw YT, de Graaf PW. CT prediction of irresectability in esophageal carcinoma: value of additional patient positions and relation to patient outcome. Abdom Imaging. 1997 Mar-Apr;22(2):132-7. doi: 10.1007/s002619900157. PMID 9013520
- [Background] Tsujimoto H, Ichikura T, Aiko S, Yaguchi Y, Kumano I, Takahata R, Matsumoto Y, Yoshida K, Ono S, Yamamoto J, Hase K. Multidetector-computed tomography attenuation values between the tumor and aortic wall in response to induction therapy for esophageal cancer and its predictive value for aortic invasion. Exp Ther Med. 2012 Feb;3(2):243-248. doi: 10.3892/etm.2011.386. Epub 2011 Nov 22. PMID 22969876
- [Background] Crehange G, Bosset M, Lorchel F, Buffet-Miny J, Dumas JL, Mercier M, Puyraveau M, Maingon P, Bosset JF. Tumor volume as outcome determinant in patients treated with chemoradiation for locally advanced esophageal cancer. Am J Clin Oncol. 2006 Dec;29(6):583-7. doi: 10.1097/01.coc.0000242346.25229.48. PMID 17148995